CLINICAL TRIAL: NCT03139266
Title: Project UPLIFT to Reduce Anxiety and Depression in CF Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: University of Michigan (Other); Boston Children's Hospital (Other); University at Buffalo (Other); Emory University (Other); Children's Hospital Medical Center, Cincinnati (Other); Johns Hopkins University (Other); Cystic Fibrosis Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HM20002923; SCHECH15A0 (Other Grant/Funding Number: Cystic Fibrosis Foundation)
Record Dates: First submitted 2017-04-24; First posted 2017-05-03 (Actual); Last update posted 2023-06-06 (Actual); Status verified 2023-06

CONDITIONS: Cystic Fibrosis; Anxiety; Depression
Keywords: cystic fibrosis; mindfulness; cognitive behavioral therapy; UPLIFT; anxiety; depression; web based intervention
MeSH Terms: conditions — Cystic Fibrosis; Anxiety Disorders; Depression | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- UPLIFT (Experimental): The Project UPLIFT intervention was designed for delivery to groups of six to eight people by telephone or Internet, though for this study the intervention will be web based only. The telephone intervention comprised eight hour-long sessions, each including check-in, instruction, skill building, and discussion, with homework between sessions. The Web intervention contains the same elements: check-in, video instruction, skill building, a discussion board, and homework between sessions. Instruction focuses on increasing knowledge about depression, cystic fibrosis (CF), cognitive behavioral therapy (CBT), and mindfulness and skills related to CBT and mindfulness.
  Interventions: Behavioral: UPLIFT
- Control Group (Other): Treatment-as-usual
  Interventions: Behavioral: Treatment as usual

INTERVENTIONS:
Behavioral: UPLIFT — Participation in the sessions involves skills practice, discussions, and group exercises based on the sessions' main topics. CBT-related topics include thought monitoring, identifying cognitive distortions, self-esteem, problem identification, goal setting, and identifying supports. Relaxation exercises, including a body scan (i.e., a mindfulness exercise) and progressive muscle relaxation, are also used for coping and to facilitate awareness of the body. Mindfulness activities include attention to skin, sights, and sounds and other meditations. Participants will practice their skills between sessions through homework assignments including monitoring and changing thoughts, and practicing relaxation exercises, meditation exercises, and mindfulness.
  Arms: UPLIFT
Behavioral: Treatment as usual — The control group will receive the recommendation to consider maintaining mental health services
  Arms: Control Group

SUMMARY:
People with CF have elevated rates of anxiety and depression when compared to the general population. Anxiety and depression can have a negative impact on adherence and disease self-management, leading to worse CF health outcomes such as respiratory symptoms, functional capacity, and health-related quality of life (HRQOL).

Project UPLIFT is a group mental health intervention that can be delivered by telephone or Web, though for this study the intervention will be web based only. Project UPLIFT was originally developed as a depression treatment and prevention program for people with epilepsy and was shown to be effective in reducing depression and increasing knowledge and skills. Recently, Project UPLIFT was revised to help people with CF manage their depression and anxiety and shown to be apparently successful in a pilot study that included adolescents and adults with CF.

The goals of this project are to determine the effectiveness of Project UPLIFT in reducing anxiety and depression in adolescents and adults with CF, as well as increasing their quality of life and other physical health-related disease outcomes.

DETAILED DESCRIPTION:
The Project UPLIFT intervention was designed for delivery to groups of six to eight people by telephone or Internet, though for this study the intervention will be web based only. The telephone intervention comprised eight hour-long sessions, each including check-in, instruction, skill building, and discussion, with homework between sessions. The Web intervention contains the same elements: check-in, video instruction, skill building, a discussion board, and homework between sessions. Instruction focuses on increasing knowledge about depression, CF, CBT, and mindfulness and skills related to CBT and mindfulness. Participation in the sessions involves skills practice, discussions, and group exercises based on the sessions' main topics. CBT-related topics include thought monitoring, identifying cognitive distortions, self-esteem, problem identification, goal setting, and identifying supports. Relaxation exercises, including a body scan (i.e., a mindfulness exercise) and progressive muscle relaxation, are also used for coping and to facilitate awareness of the body. Mindfulness activities include attention to skin, sights, and sounds and other meditations. Participants will practice their skills between sessions through homework assignments including monitoring and changing thoughts, and practicing relaxation exercises, meditation exercises, and mindfulness. A week's homework is discussed at the beginning of the next session. The program is designed to guide participants from noticing, challenging, and changing thoughts (CBT components), to staying in the present moment with acceptance of and nonreactivity to those thoughts (mindfulness components). All sessions will be co-facilitated by a layperson with CF and a doctoral student in psychology, supervised by a licensed clinical psychologist.

Once the subjects are recruited and enrolled, baseline assessment will take place and then they will be randomized into the intervention group or treatment-as-usual control group condition (recommendation to consider obtaining mental health services). All participants will complete questionnaires via the internet. Following the initial assessment, the groups will receive their assigned intervention (or control treatment) and there will be questionnaire based testing of mental health, QoL, and disease management at 2 months (immediately following the group intervention), 6 months, and 12 months.

ELIGIBILITY:
*Please note that only patients who are seen by one of our participating CF clinics (listed in "locations") will be approached about UPLIFT (if eligible) during this phase of the UPLIFT project.*

Inclusion Criteria:

First, patients will have to agree to have their contact information shared with the study team in order to be eligible.

Eligibility criteria:

* have been diagnosed with CF for at least 1 year;
* score 5-14 on the GAD-7 and/or a 5-19 on the PHQ-9;
* be ≥13 years of age;
* be English speaking; and
* not have a prominent cognitive impairment.

Exclusion Criteria:

* Persons reporting active suicidal ideation on the PHQ-9 will be excluded.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2015-04-07 (Actual); Primary Completion 2022-08-02 (Actual); Study Completion 2022-08-02 (Actual)

PRIMARY OUTCOMES:
Reduce symptoms of anxiety among UPLIFT Tx Group participants. | Baseline (at 0 week), Tx End (at 8 weeks), Follow-up (at 6 months post Tx End), Extended Follow-up (at 12 months post Tx End)
  Anxiety symptoms will be assessed with the Generalized Anxiety Disorder-7 (GAD-7)
Reduce symptoms of depression among UPLIFT Tx Group participants. | Baseline (at 0 week), Tx End (at 8 weeks), Follow-up (at 6 months post Tx End), Extended Follow-up (at 12 months post Tx End)
  Depressive Symptoms will be assessed with the Patient Health Questionnaire-9 (PHQ-9).

SECONDARY OUTCOMES:
Increase quality of life among UPLIFT Tx Group participants. | Baseline (at 0 week), Tx End (at 8 weeks), Follow-up (at 6 months post Tx End), Extended Follow-up (at 12 months post Tx End)
  Quality of Life will be assessed using the Cystic Fibrosis Questionnaire-Revised (CFQ-R).
Increase satisfaction with life among UPLIFT Tx Group participants. | Baseline (at 0 week), Tx End (at 8 weeks), Follow-up (at 6 months post Tx End), Extended Follow-up (at 12 months post Tx End)
  Satisfaction with life will be measured using the Satisfaction with Life Scale.
Improve knowledge and skills regarding self-management of anxiety and depression among UPLIFT Tx Group participants. | Baseline (at 0 week), Tx End (at 8 weeks), Follow-up (at 6 months post Tx End), Extended Follow-up (at 12 months post Tx End)
  Will be assessed using an 18-item true-false measure developed during the development of Project UPLIFT.
Increase self-efficacy among UPLIFT Tx Group participants. | Baseline (at 0 week), Tx End (at 8 weeks), Follow-up (at 6 months post Tx End), Extended Follow-up (at 12 months post Tx End)
  We will measure this using the Depression Coping Self-Efficacy Scale (DCSES).

OTHER OUTCOMES:
(Exploratory) Change in CF disease severity status. | Baseline (at 0 week), Tx End (at 8 weeks), Follow-up (at 6 months post Tx End), Extended Follow-up (at 12 months post Tx End)
  CF disease related measures will be collected from routine clinic visits that occur from the time of enrollment to final UPLIFT follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Michael S Schechter, MD, MPH, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Informed Consent Form: Parental consent (2020-04-23): https://cdn.clinicaltrials.gov/large-docs/66/NCT03139266/ICF_000.pdf
  • Informed Consent Form: Adult consent (2020-04-23): https://cdn.clinicaltrials.gov/large-docs/66/NCT03139266/ICF_001.pdf